CLINICAL TRIAL: NCT04388917
Title: Does the Use of Hemostatic Clips During the Tumor Resection Step Reduce Blood Loss During Robot-assisted Partial Nephrectomy?
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 20Urobase02
Record Dates: First submitted 2020-05-12; First posted 2020-05-14 (Actual); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: Renal Cancer; Kidney Cancer; Blood Loss
Keywords: robot assisted partial nephrectomy; tips
MeSH Terms: conditions — Kidney Neoplasms; Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Renal tumor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Clip Group: Use of Hemo-lock hemostatic clips during tumor resection to prevent bleeding
  Interventions: Procedure: Patial nephrectomy
- No Clip group: No Hemo-lock hemostatic clips used during tumor resection
  Interventions: Procedure: Patial nephrectomy

INTERVENTIONS:
Procedure: Patial nephrectomy — Partial nephrectomy assisted with robot to remove kidney cancer

SUMMARY:
One challenge of robot-assisted partial nephrectomy (RAPN) is to reduce operative blood loss. Partial nephrectomy (PN) is a complex surgery that is being made easier by robotic assistance. In this study, we determined whether the use of hemostatic clips during the tumor resection step reduced blood loss during robot-assisted partial nephrectomy. Methods: In this retrospective study, we included all consecutive patients who underwent RAPN in our university hospital from 2017 to 2019. Three experienced surgeons performed the surgery. One surgeon used Hemo-lock hemostatic clips during tumor resection to prevent bleeding, and two did not. Blood loss in the two groups was compared as the primary endpoint. The duration of clamping, operative time, complications, surgical margins, transfusions, serum creatinine and hemoglobin were compared as secondary endpoints. Results: 53 patients were included, 36 in the No-clip group and 17 in the Clip group. Our two groups were comparable for age, weight, Charlson score, tumor size and RENAL score. There was a significant difference between the two groups for median blood loss 50 mL in the Clip group versus 300 mL in the No-clip group (p = 0.0001), whereas median operating time was shorter in the No-clip group, 140 min versus 180 min for the Clip group (p = 0.044). No other criterion showed a significant difference. The use of Hemo-lock during the tumor resection step in RAPN reduced blood loss without impairing renal function. Larger studies are still needed to confirm our findings.

ELIGIBILITY:
Inclusion Criteria:

* all consecutive patients who underwent Robot Assisted Partial Nephrectomy

Exclusion Criteria:

* patient off clamping or partial clamping

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all consecutive patients who underwent Robot Assisted Partial Nephrectomy
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Blood loss in the two groups was compared | 3 years
  It was mesured during the surgery by amount of blood drawn

SECONDARY OUTCOMES:
operative time | 3 years
  duration from the begining to the end of the surgery
duration of clamping | 3 years
  time between the clips set and remove during the surgery for patient of clip group
incidence of complications | 3 years
  rate of complication after surgery

IPD SHARING:
Plan to Share IPD: No
no data sharing plan has been established